CLINICAL TRIAL: NCT01516736
Title: Pivotal Study in Breast Cancer Patients Investigating Efficacy and Safety of LA-EP2006 and Neulasta®
Brief Title: Phase III Study Comparing the Efficacy and Safety of LA-EP2006 and Peg-Filgrastim
Acronym: PROTECT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Sandoz GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LA-EP06-302
Record Dates: First submitted 2012-01-13; First posted 2012-01-25 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Chemotherapy-induced Neutropenia; Breast Cancer
Keywords: Pegfilgrastim; G-CSF; neutropenia; breast cancer; myelosuppressive chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LA-EP2006 (Experimental): During each chemotherapy cycle eligible patients receive LA-EP2006 s.c. post chemotherapy application.
  Interventions: Drug: LA-EP2006
- Neulasta® (Active Comparator): During each chemotherapy cycle eligible patients receive Neulasta® s.c. post chemotherapy application.
  Interventions: Drug: Neulasta®

INTERVENTIONS:
Drug: LA-EP2006 — Eligible patients are scheduled to receive six cycles of chemotherapy every three weeks. During each chemotherapy cycle LA-EP2006 is injected s.c. post chemotherapy application.
  Other Names: pegfilgrastim
  Arms: LA-EP2006
Drug: Neulasta® — Eligible patients are scheduled to receive six cycles of chemotherapy every three weeks. During each chemotherapy cycle Neulasta® is injected s.c. post chemotherapy application.
  Other Names: pegfilgrastim; Neulasta
  Arms: Neulasta®

SUMMARY:
The study will assess the efficacy of LA-EP2006 compared to Neulasta® with respect to the mean duration of severe neutropenia during treatment with myelosuppressive chemotherapy in breast cancer patients.

DETAILED DESCRIPTION:
The Pegfilgrastim Randomized Oncology (Supportive Care) Trial to Evaluate Comparative Treatment (PROTECT-2) was a confirmatory efficacy and safety study designed to compare the proposed biosimilar LA-EP2006 with the reference pegfilgrastim in woman with early stage breast cancer receiving (neo)-adjuvant myelosuppressive chemotherapy. Patient received TAC (intravenous docetaxel 75mg/m^2, doxorubicin 50 mg/m^2, and cyclophosphamide 500mg/m^2) on day1 of each cycle, for six or more cycles. A total of 308 patients were randomized to LA-EP2006 (n=155) or reference Neulasta® (n=153). Treatment was given subcutaneously on day 2 of each cycle. The primary end point was the duration of severe neutropenia (DSN) during Cycle 1 (defined as number of consecutive days with absolute neutrophil count <0.5 × 10^9 cells/L). LA-EP2006 was equivalent to the reference product in DSN (difference: -0.16 days; 95% CI [-0.40, 0.08]). Further, LA-EP2006 and the reference pegfilgrastim showed no clinically meaningful differences regarding efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven breast cancer
* eligible for six cycles of neoadjuvant or adjuvant chemotherapy

Exclusion Criteria:

* concurrent or prior chemotherapy for breast cancer
* concurrent or prior anti-cancer treatment for breast cancer such as endocrine therapy, immunotherapy, monoclonal antibodies, and/or biological therapy
* concurrent prophylactic antibiotics
* previous therapy with any G-CSF (granulocyte-colony stimulating factor) product

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz Biopharmaceutical Clinical Development, Study Chair — Sandoz Biopharmaceuticals
Locations (47):
- United States (10):
  - Sandoz Investigational Site, Hot Springs, Arkansas
  - Sandoz Investigational Site, Jonesboro, Arkansas
  - Sandoz Investigational Site, Corona, California
  - Sandoz Investigational Site, Wichita, Kansas
  - Sandoz Investigational Site, Mount Sterling, Kentucky
  - Sandoz Investigational Site, Detroit, Michigan
  - Sandoz Investigational Site, Bismarck, North Dakota
  - Sandoz Investigational Site, Eugene, Oregon
  - Sandoz Investigational Site, Germantown, Tennessee
  - Sandoz Investigational Site, Newport News, Virginia
- Sandoz Investigational Site, San Miguel de Tucumán, Argentina
- Sandoz Investigational Site, Temuco, Chile
- India (14):
  - Sandoz Investigational Site, Chennai
  - Sandoz Investigational Site, Delhi
  - Sandoz Investigational Site, Gujarat
  - Sandoz Investigational Site, Hyderabad
  - Sandoz Investigational Site, Karamsad
  - Sandoz Investigational Site, Lucknow
  - Sandoz Investigational Site, Maharashtra
  - Sandoz Investigational Site, Mangalore
  - Sandoz Investigational Site, Mumbai
  - Sandoz Investigational Site, Pradesh
  - Sandoz Investigational Site, Surat
  - Sandoz Investigational Site, Vadodara
  - Sandoz Investigational Site, Vellore
  - Sandoz Investigational Site, Visakhapatnam
- Malaysia (3):
  - Sandoz Investigational Site, George Town
  - Sandoz Investigational Site, Kampung Baharu Nilai
  - Sandoz Investigational Site, Kelantan
- Sandoz Investigational Site, San Juan, Puerto Rico
- Russia (13):
  - Sandoz Investigational Site, Arkhangelsk
  - Sandoz Investigational Site, Bashkortostan
  - Sandoz Investigational Site, Bryansk
  - Sandoz Investigational Site, Kazan'
  - Sandoz Investigational Site, Krasnoyarsk
  - Sandoz Investigational Site, Moscow
  - Sandoz Investigational Site, Omsk
  - Sandoz Investigational Site, Orenburg
  - Sandoz Investigational Site, Oryol
  - Sandoz Investigational Site, Rostov-on-Don
  - Sandoz Investigational Site, Saint Petersburg
  - Sandoz Investigational Site, Tomsk
  - Sandoz Investigational Site, Vladimir
- Spain (4):
  - Sandoz Investigational Site, Barcelona
  - Sandoz Investigational Site, Madrid
  - Sandoz Investigational Site, Santiago de Compostela
  - Sandoz Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blackwell K, Donskih R, Jones CM, Nixon A, Vidal MJ, Nakov R, Singh P, Schaffar G, Gascon P, Harbeck N. A Comparison of Proposed Biosimilar LA-EP2006 and Reference Pegfilgrastim for the Prevention of Neutropenia in Patients With Early-Stage Breast Cancer Receiving Myelosuppressive Adjuvant or Neoadjuvant Chemotherapy: Pegfilgrastim Randomized Oncology (Supportive Care) Trial to Evaluate Comparative Treatment (PROTECT-2), a Phase III, Randomized, Double-Blind Trial. Oncologist. 2016 Jul;21(7):789-94. doi: 10.1634/theoncologist.2016-0011. Epub 2016 Apr 18. PMID 27091420
- [Derived] Blackwell K, Gascon P, Jones CM, Nixon A, Krendyukov A, Nakov R, Li Y, Harbeck N. Pooled analysis of two randomized, double-blind trials comparing proposed biosimilar LA-EP2006 with reference pegfilgrastim in breast cancer. Ann Oncol. 2017 Sep 1;28(9):2272-2277. doi: 10.1093/annonc/mdx303. PMID 28637287

RESULTS

PARTICIPANT FLOW:
Groups:
- Neulasta®: During each chemotherapy cycle eligible patients receive Neulasta® s.c. post chemotherapy application.
  Neulasta®: Eligible patients are scheduled to receive six cycles of chemotherapy every three weeks. During each chemotherapy cycle pegfilgrastim is injected s.c. post chemotherapy application.
Period: Overall Study
Arm/Group | LA-EP2006 | Neulasta®
Started (FAS/SAF full analysis set and safety analysis set) | 155 | 153
Completed (1 more patient, Neulasta arm died but been withdrawn earlier, not included in participant flow-death) | 135 | 140
Not Completed | 20 | 13
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Adverse Event | 4 | 5
Not completed — Death | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Other (not specified) | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patient demographics (FAS set)
Groups:
- Total: Total of all reporting groups
Arm/Group | LA-EP2006 | Neulasta® | Total
Number analyzed (Participants) | 155 | 153 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (10.50) | 49.1 (10.07) | 48.9 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 153 | 308
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 145 | 147 | 292
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The 2 patients with race "More than one race" were reported as Hispanic origin.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 62 | 58 | 120
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 2 | 3
    White | 90 | 93 | 183
    More than one race | 2 | 0 | 2
    Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.56 (5.771) | 26.49 (5.126) | 26.53 (5.450)
Time since diagnosis [Median (Full Range); unit: months] — Population: For 2 patients in the Neulasta treatment group, the date of initial diagnosis was incomplete.
  months
    number analyzed (Participants) | 155 | 151 | 306
    (all) | 1.28 [0.2 to 42.3] | 1.28 [0.3 to 11.2] | 1.28 [0.2 to 42.3]
Disease stage [Count of Participants; unit: Participants] — TNM Disease stage was defined according to the American Joint Committee on Cancer (AJCC): (I) = T1 N0 M0 / T0 N1mi M0 / T1 N1mi M0; (II) = T0 N1 M0 / T1 N1 M0 / T2 N0 M0 / T2 N1 M0 / T3 N0 M0; (III) = T0 N2 M0 / T1 N2 M0 / T2 N2 M0 / T3 N1 M0 / T3 N2 M0 / T4 N0 M0 / T4 N1 M0 / T4 N2 M0 / AnyT N3 M0; (IV) = AnyT AnyN M1; T: size or direct extent of the primary tumour; N: degree of spread to regional lymph nodes; N1mi: Micrometastases (> 0.2 mm and/or > 200 cells, but none > 2.0 mm); M: presence of distant; https://www.cancer.gov/types/breast/hp/breast-treatment-pdq#link/_27
  Participants
    I | 7 | 13 | 20
    II | 70 | 61 | 131
    III | 78 | 78 | 156
    IV | 0 | 1 | 1
Previous breast cancer surgery [Count of Participants; unit: Participants] | 154 | 152 | 306
Previous radiotherapy [Count of Participants; unit: Participants] | 2 | 1 | 3
ECOG performance status [Count of Participants; unit: Participants] — Grading according to ECOG:
  0: Fully active, able to carry on all pre-disease performance without restriction 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work 2: Ambulatory and capable of all self-care but unable to carry out any work activities up and about more than 50% of waking hours 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  Participants
    0 | 117 | 110 | 227
    1 | 36 | 43 | 79
    2 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Duration of Severe Neutropenia (DSN) During Cycle 1 of Chemotherapy
Description: Mean duration of severe neutropenia, defined as number of consecutive days with ANC <0.5 × 10^9/l (grade 4 neutropenia).
Time Frame: 21 days (Cycle 1 of chemotherapy treatment)
Population: Missing patients in FAS set due to blind data review meeting decision (no ANC profiles available). FAS set = full analysis set; PP set = per protocol set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 155 | 153
days
  FAS: number analyzed (Participants) | 151 | 149
  FAS | 1.36 (1.133) | 1.19 (0.984)
  PP: number analyzed (Participants) | 148 | 144
  PP | 1.34 (1.141) | 1.19 (0.991)
Statistical Analysis 1: Comparison: LA-EP2006 vs Neulasta®; The primary objective of the study was to compare LA-EP2006 and Neulasta in terms of the DSN in Cycle 1. It was to be shown in a hierarchical way: 1. that LA-EP2006 is equivalent (margin: ±1 day) to Neulasta® with respect to DSN duration in Cycle 1 and, if this was successfully established, 2. that LA-EP2006 is non-inferior (margin: -0.6 days) to Neulasta® with respect to DSN duration in Cycle 1; Test type: Equivalence — The testing procedure was set up in a hierarchical structure, where first equivalence between LA-EP2006 and Neulasta® was assessed (margin ±1 day) and only if this was successfully established, non-inferiority between the two products was tested using a tighter margin of -0.6 days; p = 0.05, ANCOVA; The primary endpoints was analyzed with analysis of covariance (ANCOVA); Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.40 to 0.08]
Statistical Analysis 2: Comparison: LA-EP2006 vs Neulasta®; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, ANCOVA; The primary endpoints was analyzed with analysis of covariance (ANCOVA); Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.40 to 0.08]

2. Secondary Outcome: Incidence of Febrile Neutropenia (FN)
Description: FN was defined as oral temperature ≥ 38.3°C while having an absolute neutrophil count (ANC) < 0.5 × 10^9 cells/L. Serious treatment-emergent adverse events (TEAEs) were reconciled with the fever and ANC results recorded in the patient diary and CRF and therefore only the serious TEAEs of FN ("febrile neutropenia", "neutropenic sepsis") were taken into account.
Time Frame: across all cycles (18 weeks)
Population: FAS set = full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 155 | 153
Participants
  Cycle 1 | 12 | 15
  Cycle 2 | 0 | 3
  Cycle 3 | 3 | 1
  Cycle 4 | 2 | 1
  Cycle 5 | 0 | 1
  Cycle 6 | 2 | 1
  All cycles (at least on incidence) | 16 | 20

3. Secondary Outcome: Number of Patients With at Least One Episode of Fever by Cycle and Across All Cycles
Description: Fever was defined as an oral body temperature of ≥ 38.3°C. Fever episodes were described by maximum oral temperature and the number of patients who had fever at least once.
Time Frame: across al cycles (18 weeks)
Population: Patients with more than 1 event during the study (overall) are counted only once. FAS set = full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 155 | 153
Participants
  Cycle 1 | 13 | 17
  Cycle 2 | 8 | 6
  Cycle 3 | 4 | 7
  Cycle 4 | 5 | 10
  Cycle 5 | 3 | 3
  Cycle 6 | 5 | 4
  Overall | 32 | 35

4. Secondary Outcome: Depth of ANC Nadir in Cycle 1
Description: The depth of ANC nadir was defined as the patient's lowest ANC (10^9 cells/L) in Cycle 1.
Time Frame: Cycle 1 (3 weeks)
Population: FAS set = full analysis set
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 152 | 149
10^9 cells/L | 0.490 (0.7205) | 0.444 (0.5684)

5. Secondary Outcome: Number of Patients With ANC Nadir Per Day in Cycle 1
Description: Numbers of patients with ANC nadir based per day during Cycle 1 are given.
Time Frame: Cycle 1 (3 weeks)
Population: FAS set = full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 155 | 153
Participants
  Days 1-5 | 1 | 0
  Day 6 | 9 | 8
  Day 7 | 117 | 109
  Day 8 | 20 | 30
  Day 9 | 3 | 2
  Days 10-15 | 2 | 0
  not definable | 3 | 4

6. Secondary Outcome: Time to ANC Recovery in Days in Cycle 1
Description: Time to absolute neutrophil count (ANC) recovery was defined as the time in days from ANC nadir until the patient's ANC had increased to ≥ 2 × 10^9 cells/L after the nadir in Cycle 1.
Time Frame: across Cycle 1 (3 weeks)
Population: FAS set = full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 155 | 153
days | 2.11 (0.889) | 2.04 (0.951)

7. Secondary Outcome: Frequency of Infections by Cycle and Across All Cycles
Description: The number of patients with infections was recorded for each cycle and across all cycles. Infections were identified by the AE documentation page selecting all events coded with System Organ Class "Infections and Infestations".
Time Frame: across all cycles (18 weeks)
Population: Patients with more than 1 event during the study (overall) are counted only once. FAS set = full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 155 | 153
Participants
  Cycle 1 | 10 | 14
  Cycle 2 | 5 | 3
  Cycle 3 | 2 | 5
  Cycle 4 | 4 | 5
  Cycle 5 | 2 | 6
  Cycle 6 | 5 | 5
  Overall | 26 | 32

8. Secondary Outcome: Mortality Due to Infection
Description: Number of patients with death due to infections
Time Frame: Study course (19 weeks)
Population: FAS set = full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 155 | 153
Participants
  Yes | 0 | 0
  No | 155 | 153

ADVERSE EVENTS:
Time Frame: Patients were followed for a 4-week safety period from the last administration of pegfilgrastim.
Description: Severity of treatment-emergent adverse events (TEAEs) was captured by CTCAE (Common Toxicology Criteria for Adverse Events) grading. SAF set = safety analysis set was used
Arm/Group | LA-EP2006 | Neulasta®
All-Cause Mortality (participants affected / at risk) | 3/155 | 2/153
Serious Adverse Events (participants affected / at risk) | 29/155 | 32/153
Other Adverse Events (participants affected / at risk) | 147/155 | 144/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LA-EP2006 (N=155) | Neulasta® (N=153)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 19
Neutropenia (Blood and lymphatic system disorders) | 4 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 5
Diarrhea (Gastrointestinal disorders) | 2 | 5
Vomiting (Gastrointestinal disorders) | 2 | 4
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Asthenia (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Pericardial hemorrhage (Cardiac disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Shock hemorrhagic (Vascular disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 1
Hepatic hemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal hemorrhage (Renal and urinary disorders) | 1 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LA-EP2006 (N=155) | Neulasta® (N=153)
Gastrointestinal disorders (Gastrointestinal disorders) | 111 | 100
General disorders and administration site conditions (General disorders) | 93 | 90
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 77 | 72
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 79 | 71
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 45 | 40
Nervous system disorders (Nervous system disorders) | 32 | 25
Infections and infestations (Infections and infestations) | 24 | 27
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 21 | 18
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 14 | 21
Investigations (Investigations) | 17 | 14
Vascular disorders (Vascular disorders) | 14 | 8
Reproductive system and breast disorders (Reproductive system and breast disorders) | 10 | 5
Eye disorders (Eye disorders) | 8 | 6
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 | 5
Renal and urinary disorders (Renal and urinary disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes